CLINICAL TRIAL: NCT05957120
Title: Subclinical Impairment of Cardiovascular System in Patients With Psoriasis
Acronym: PaS
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Eva Klara Merzel Šabović, Eva Klara Merzel Šabović, MD, University Medical Centre Ljubljana
Other Study IDs: PICANTI
Record Dates: First submitted 2023-06-18; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Psoriasis; Inflammation; Endothelial Dysfunction; Metabolic Disturbance; Insulin Resistance; Coagulation Disorder; Thrombocyte Disorders
Keywords: Psoriasis; Endothelial dysfunction; Inflammation; Insulin resistance; Biologic therapy
MeSH Terms: conditions — Psoriasis; Inflammation; Insulin Resistance; Hemostatic Disorders; Blood Platelet Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Withdrawal of blood for laboratory analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients on local therapy: 20 patients on local antipsoriatic therapy (either corticosteroid cream/ointment, calcipotriol or combination (corticosteroid and calcipotriol); duration of treatment varies in cohort of patients
- Patients on methotrexate: 20 patients on methotrexate with dosage adjusted by weight; duration of treatment varies in cohort of patients
- Patients on biologic therapy with anti-tumor necrosis factor-alpha: 20 patients on adalimumab - 40 mg every two weeks (or 40 mg weekly if the response was previously insufficient); duration of treatment varies in cohort of patients
- Patients on biologic therapy with anti-interleukin-17: 20 patients on secukinumab - 300 mg monthly (or 300 mg every two weeks if the response was previously insufficient); duration of treatment varies in cohort of patients
- Patients on biologic therapy with anti-interleukin-23: 20 patients on guselkumab - 100 mg every 8 weeks; duration of treatment varies in cohort of patients
- Controls: 20 subjects who are age-matched

SUMMARY:
A cross-sectional study will be conducted, which will include 80 young patients with psoriasis, aged 30-45 years, treated with five different types of antipsoriatic treatment, and 20 healthy patients. All 100 subjects will be subjected to anthropometric measurements, blood will be collected for laboratory tests, and an imaging test will be performed to determine the function of the endothelium and arterial stiffness. The results will then be statistically analyzed.

DETAILED DESCRIPTION:
Research design: A cross-sectional study will be conducted, which will include 80 young patients with psoriasis, aged 30-45 years, without other chronic diseases, treated with five different types of treatment (local therapy, methotrexate, inhibitor of tumor necrosis factor α, inhibitor of interleukin 17 and inhibitor of interleukin 23), and 20 healthy patients aged 30-45 years. All 100 subjects will be subjected to anthropometric measurements (measurement of weight, height, systolic and diastolic blood pressure, heart rate, waist circumference), blood will be collected for laboratory tests (full blood count with differential, CRP, serum electrolytes, lipid panel, fasting glucose, HbA1c, alanine aminotransferase, aspartate aminotransferase, creatinine, urea, TNF-alpha, IL-6, IL-12, IL-17, IL-23, hsCRP, IFN-gamma, TRANCE, TRAIL, GDF-15, D-dimer, fibrinogen, overall haemostasis potential, overall coagulation potential, VCAM-1, ECAMs), and an imaging test (flow-mediated dilation and measurement of pulse wave velocity) will be performed to determine the function of the endothelium and arterial stiffness. The results will then be statistically analyzed.

Aim of the study: The impact of chronic systemic inflammation in psoriasis on subclinical defects in the cardiovascular system (endothelial dysfunction, arterial stiffness, insulin resistance, platelet activation, and coagulation activation) and their effects on each other will be studied. In addition, the effect of the five main types of psoriasis treatment on all listed subclinical defects of the cardiovascular system will be investigated. Moreover, it will be investigated whether the type of treatment affects systemic inflammation in psoriasis in the same manner.

Expected results: It is expected that all five groups of patients will differ from each other in terms of the degree of subclinical impairment of the cardiovascular system, depending on the expression of psoriasis and the type of treatment they receive. This will form the basis for establishing preventive measures against cardiovascular diseases in patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

- patients with psoriasis aged 30 to 45 years in stable phase of the disease for at least last 6 months

Exclusion Criteria:

* any treatment besides treatment of psoriasis
* carotid disease
* heart failure
* atrial fibrillation
* diabetes type 1 or 2
* cardiovascular event in the past
* chronic kidney disease stage 3, 4, 5 or end-stage kidney disease
* psoriatic arthritis or any other rheumatic disease
* malignancy
* menopause in women
* other chronic inflammatory diseases

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 5 groups of patients with psoriasis that are treated in our hospital with either local treatment, methotrexate, adalimumab, secukinumab or guselkumab will be included in the study. Included patients will be aged 30 to 45 years and will be without other chronic disease besides psoriasis and without other treatment besides antipsoriatic treatment to investigate the isolated effect of psoriasis on observed parameters (endothelial function, endothelial activation, inflammation, insulin resistance, metabolic disturbances, activation of coagulation and activation of platelets).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Arterial function - endothelial function | through study completion, an average of 6 months
  Endothelial function (flow-mediated dilation)
Arterial function - arterial stiffness | through study completion, an average of 6 months
  Arterial stiffness (pulse wave velocity)
Endothelial activation | through study completion, an average of 6 months
  Circulating markers of endothelial activation (E-selectin, vascular cell adhesion molecule-1 (VCAM-1), Endothelial cell adhesion molecules (ECAMs))

SECONDARY OUTCOMES:
Inflammation | through study completion, an average of 6 months
  Circulating markers of inflammation (tumor necrosis factor-alpha (TNF-alpha), interleukin (IL)-6, IL-12, IL-17, IL-23, high sensitivity C-reactive protein (hs-CRP), interferon-gamma, TNF-related activation-inducing ligand (TRANCE), TNF-related apoptosis-inducing ligand (TRAIL), Growth/differentiation factor-15 (GDF-15), neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR))
Insulin resistance | through study completion, an average of 6 months
  Circulating markers of insulin resistance (fasting glucose, insulin), HOMA-IR equation (Homeostatic Model Assessment for Insulin Resistance)
Metabolic disturbances - dyslipidemia | through study completion, an average of 6 months
  Parameters of (pre)metabolic syndrome (lipid panel)
Metabolic disturbances | through study completion, an average of 6 months
  Parameters of (pre)metabolic syndrome (TyG (triglyceride-glucose index))
Liver steatosis | through study completion, an average of 6 months
  Laboratory markers (aspartate aminotransferase (AST), Alanine Aminotransferase (ALT), Fib4 score (Fibrosis-4))
Coagulation | through study completion, an average of 6 months
  Circulating markers of coagulation activation (D-dimer, fibrinogen)
Activation of hemostasis | through study completion, an average of 6 months
  Hemostatic assay (overall hemostasis potential (OHP) assay)
Activation of coagulation | through study completion, an average of 6 months
  Coagulation assay (overall coagulation potential (OCP) assay)
Platelet activation (1) | through study completion, an average of 6 months
  Circulating markers of platelet activation (mean platelet volume (MPV)
Platelet activation (2) | through study completion, an average of 6 months
  Circulating markers of platelet activation (P-selectin)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Klara Merzel Sabovic, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Merzel Sabovic EK, Kraner Sumenjak T, Bozic Mijovski M, Janic M. Residual non-specific and disease-specific inflammatory markers in successfully treated young psoriasis patients: a cross-sectional study. Immunol Res. 2025 Jan 8;73(1):28. doi: 10.1007/s12026-024-09584-4. PMID 39775226
- [Derived] Merzel Sabovic EK, Kraner Sumenjak T, Bozic Mijovski M, Janic M. Arterial function is preserved in successfully treated patients with psoriasis vulgaris. Sci Prog. 2024 Oct-Dec;107(4):368504241287893. doi: 10.1177/00368504241287893. PMID 39403781
- [Derived] Merzel Sabovic EK, Kraner Sumenjak T, Janic M. Residual metabolic burden in young psoriasis patients successfully treated with biologics. Arch Dermatol Res. 2024 Sep 27;316(9):647. doi: 10.1007/s00403-024-03403-4. PMID 39331218